CLINICAL TRIAL: NCT01654341
Title: A RANDOMIZED CLINICAL TRIAL TO EVALUATE THE EFFECTIVENESS OF A MULTI-MODAL INTERVENTION IN FRAIL AND PREFRAIL OLDER PEOPLE WITH TYPE 2 DIABETES ON FRAILTY AND QUALITY OF LIFE: THE MID-Frail STUDY
Brief Title: Multi-Modal Intervention In Frail And Prefrail Older People With Type 2 Diabetes
Acronym: MID-Frail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Getafe (Other)
Collaborators: Cardiff University (Other); Igen Biotech SL (Unknown); University Hospital, Bordeaux (Other); Hexabio Sarl (Unknown); University of Campania Luigi Vanvitelli (Other); University Hospital, Toulouse (Other); University of Ulm (Other); University Ghent (Other); University of Castilla-La Mancha (Other); Univerzita Karlova v Praze (Other); Niche Science & Technology Ltd (Unknown); Catholic University of the Sacred Heart (Other); Vrije Universiteit Brussel (Other); Diabetes Frail Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MID-Frail; 278803-2 (Other: European Commission: CORDIS: Seventh Framework Programme (FP7)); NCT01541787 (obsolete NCT alias)
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exercise; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care Group (No Intervention): Subjects undergo usual standard of care
- Intervention Group (Experimental): Intervention with exercise, dietary and educational programs
  Interventions: Behavioral: Exercise, dietary and educational program

INTERVENTIONS:
Behavioral: Exercise, dietary and educational program
  Arms: Intervention Group

SUMMARY:
The MID-Frail STUDY project focuses on the use of interventions designed to improve functional status and enhance quality of life (rather than traditional treatments such as glucose- and blood pressure- lowering) by acting on the mechanisms involved in producing frailty and its progression to adverse outcomes.

DETAILED DESCRIPTION:
Detailed Description: Subjects enrolled in the main study will also be invited to join the following sub-studies:

GENEFRAIL: this sub-study aims to determine the polymorphisms of several genes associated to frailty, in order to establish its predictive value for developing disability and response to treatment as well METABOFRAIL: this sub-study aims to investigate the metabolomic profile of frail and pre-frail patients. SARTRAIN: the combination of the assessment tools used in SARTRAIN (ARFI US, MRI, posturographic measurements) will provide a comprehensive study of the structural and functional characteristics of muscle and adjacent tissues and their change with time and the intervention. MID- POW: this sub-study aims to investigate changes in muscle power.

The project also include an randomized controlled ancillary study: SENSOLE for which the aim is to investigate the potential effects of vibrating insoles device on gait and posture.

ELIGIBILITY:
Inclusion criteria:

* Participant is willing and able to give written informed consent for participation in the study.
* Subjects aged 70 years or older, with a diagnosis of type 2 diabetes mellitus for at least 2 years.
* Require to fulfill Fried ́s criteria for frail or pre-frail individuals.

Exclusion criteria:

* Barthel score lower than 60 points.
* Inability to carry out SPPB test (total score=0).
* Mini Mental State Examination score less than 20 points.
* Subjects unwilling or unable to consent or unable to participate safely in intervention program.
* Previous history of myocardial infarction within 6 months, unstable angina or congestive heart failure in III-IV NYHA stage.
* Clinically instable patients in the clinical judgment of the investigator.
* Terminal illness (life expectancy < 6 months).
* Any other condition that, in the clinical judgment of the investigator, means that it would not in the patient's best interests to enter the study.
* Current participation in clinical trial or any other investigational study.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 986 (Actual)
Dates: Start 2013-12; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Changes in summary ordinal score on the Short Physical Performance Battery test | 2 years
  The Short Physical Performance Battery (SPPB) is a simple test to measure lower extremity function using tasks that mimic daily activities. The SPPB examines 3 areas of lower extremity function; static balance, gait speed, and getting in and out of a chair. These areas represent essential tasks important for independent living and are thus an important outcome measure for patients with cardiovascular and pulmonary disease.

SECONDARY OUTCOMES:
Lawton Instrumental Activity of Daily Living (IADL) scale | 2 years
Barthel index of activities of daily living | 2 years
Euro-Quality of Life (QoL) index | 2 years
Economic costs/healthcare expenditure due to diabetes and its impact on disability and quality of life, | 2 years
  Economic costs/healthcare expenditure due to diabetes and its impact on disability and quality of life, using an economic model embracing the direct health-related costs (in-patient, out-patient, pharmaceutical, etc), formal care costs (home care, respite care, day centers, etc) and the informal care costs (carer).
Symptomatic hypoglycaemia | 2 years
  Episodes of symptomatic hypoglycaemia (i.e., a recorded blood sugar less than 4 mmol/L, or symptoms or signs attributed to low blood sugar and responding to appropriate treatment)
Hospital admissions | 2 years
  Episodes of hospital admission (i.e., any admission involving an overnight stay)
Episodes of permanent institutionalization | 2 years
  Episodes of permanent institutionalization (i.e., permanent move to any care setting other than the patient's own home, where paid staff are available to provide care if needed at any time during the day or night).
Caregiver Strain Index | 2 years
  Burden of the carer, as assessed by the modified Caregiver Strain Index
Mortality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Leocadio Rodríguez Mañas, MD, Principal Investigator — Hospital Universitario de Getafe
Locations (1):
- Hospital Universitario de Getafe, Madrid, Getafe, Spain

REFERENCES:
- [Derived] Laosa O, Topinkova E, Bourdel-Marchasson I, Vellas B, Izquierdo M, Paolisso G, Hardman T, Zeyfang A, Pedraza L, Carnicero JA, Rodriguez-Manas L, Sinclair AJ; MIDFRAIL consortium. Long-term frailty and physical performance transitions in older people with type-2 diabetes. The MIDFRAIL randomized clinical study. J Nutr Health Aging. 2025 Apr;29(4):100512. doi: 10.1016/j.jnha.2025.100512. Epub 2025 Feb 14. PMID 39954533
- [Derived] Regueme SC, Cowtan C, Sedgelmaci MY, Kelson M, Poustis J, Rodriguez-Manas L, Sinclair AJ, Dallaudiere B, Bourdel-Marchasson I. A Therapeutic Insole Device for Postural Stability in Older People With Type 2 Diabetes. A Feasibility Study (SENSOLE Part I). Front Med (Lausanne). 2019 Jun 27;6:127. doi: 10.3389/fmed.2019.00127. eCollection 2019. PMID 31316984
- [Derived] Rodriguez-Manas L, Bayer AJ, Kelly M, Zeyfang A, Izquierdo M, Laosa O, Hardman TC, Sinclair AJ, Moreira S, Cook J; MID-Frail Consortium. An evaluation of the effectiveness of a multi-modal intervention in frail and pre-frail older people with type 2 diabetes--the MID-Frail study: study protocol for a randomised controlled trial. Trials. 2014 Jan 24;15:34. doi: 10.1186/1745-6215-15-34. PMID 24456998